CLINICAL TRIAL: NCT01522833
Title: Non-Small-Cell Lung Cancer Patients Treated With Erlotinib Six Months or Longer: Demographics, Treatment and Outcome Characteristics of Patient Cases in a Community-Based Setting
Brief Title: Non Small Cell Lung Cancer Patients Treated With Erlotinib Six Months or Longer
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRI OUTCOMES 13
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSLCL; Erlotinib; Tarceva
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue-testing will be performed or test results will be reviewed to identify EGFR-wt and EGFR mutation positive advanced non small cell lung cancer (NSCLC) patient cases with an erlotinib-treatment duration of six months or longer (as 2nd/3rd line and/or maintenance single-agent therapy) in a community-based setting.
  Biopsy specimens from enrolled patient cases who are EGFR-wt will be evaluated via exploratory genetic analysis for correlated biomarkers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: EGFR Wild Type patients
- Cohort B: EGFR mutation patients

SUMMARY:
With roughly 80% of cancer patients receiving their oncology care in the community setting, the investigators are proposing to sample from a community-based center to evaluate the percentage of epidermal growth factor receptor (EGFR)-wild type patients that gain benefit from erlotinib and assess the clinical characteristics that are associated with erlotinib-responders. Additionally, biopsy specimens from enrolled patient cases that are EGFR-wt will be evaluated via exploratory genetic analysis for correlated markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had NSCLC.
* Patients must have received erlotinib (single-agent) for six months or longer for NSCLC in the second/third line setting or as maintenance therapy.
* Patients must have tissue available for EGFR-mutation status testing (if not previously performed) or EGFR-mutation status test results available.
* Patients must have tissue available for exploratory genetic analysis.
* Patients must have all clinical information, treatment response data and outcomes data available for review.
* Patients must be deceased.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EGFR-wt and EGFR mutation positive advanced NSCLC patient cases with an erlotinib-treatment duration of six months or longer (as 2nd/3rd line and/or maintenance single-agent therapy) in a community-based setting
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
demographics | 24 months
  To describe patient demographic characteristics of patients with erlotinib (single-agent) treatment duration of six months or longer, including patients who are EGFR-wt. Demographic characteristics include age, race,ethnicity, date of initial diagnosis, age at initial diagnosis, location of biopsy at diagnosis, extent of disease with description and location of metastatic sites, histology,and smoking history.
treatment characteristics | 24 months
  To describe patient treatment and characteristics of patients with erlotinib (single-agent) treatment duration of six months or longer, including patients who are EGFR-wt. Including number and kind of prior therapies, disease stage at initial diagnosis, sites of metastasis at time of erlotinib treatment, prior surgery, and radiation.
outcome characteristics | 24 months
  To describe patient outcome characteristics of patients with erlotinib (single-agent) treatment duration of six months or longer, including patients who are EGFR-wt including the reason for discontinuing erlotinib treatment, best response to erlotinib treatment and did patient receive any dose modifications while receiving erlotinib treatment.

SECONDARY OUTCOMES:
Biomarker characteristics | 24 months
  To explore biomarker (BM) characteristics of EGFR-wt erlotinib responders.
Exploratory genetic analysis | 24 months
  Biopsy specimens from enrolled patient cases who are EGFR-wt will be evaluated via exploratory genetic analysis for correlated biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States